CLINICAL TRIAL: NCT07010133
Title: Be Well at Work-Plus: A Depression and Physical Activity Intervention for Hospital Service Workers (Aim 3).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-0260; K23HL157763 (NIH)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Depression; Physical Inactivity
Keywords: Depression; Physical Activity; Employees; Worker Health; Low-income; Social needs
MeSH Terms: conditions — Depression; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a pilot randomized controlled trial with a waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention (Experimental): The intervention consists of assessment of depression and work impairment, work-focused cognitive behavioral therapy, work coaching, social needs screening and referral, and text message support for mood and physical activity.
  Interventions: Behavioral: A workplace-based depression intervention for low-wage hospital workers
- Waitlist Control (Active Comparator): Delivered after a 4-month waitlist period, the intervention consists of assessment of depression and work impairment, work-focused cognitive behavioral therapy, work coaching, social needs screening and referral, and text message support for mood and physical activity.
  Interventions: Behavioral: A workplace-based depression intervention for low-wage hospital workers

INTERVENTIONS:
Behavioral: A workplace-based depression intervention for low-wage hospital workers — This intervention is a remotely delivered workplace-based depression intervention that is tailored to the specific social and behavioral needs of low-wage hospital service workers. The intervention involves assessment of depression-related work impairment, work-focused cognitive behavioral therapy, work coaching, social needs screening and referral, and text message support for mood and physical activity.

SUMMARY:
This small randomized controlled trial will evaluate a workplace-based depression intervention that is tailored to the specific social and behavioral needs of low-wage hospital service workers. The intervention involves assessment of depression-related work impairment, work-focused cognitive behavioral therapy, work coaching, social needs screening and referral, and text message support for mood and physical activity.

DETAILED DESCRIPTION:
Depression and physical inactivity are leading contributors to cardiometabolic diseases such as obesity, diabetes, and cardiovascular disease. Low-wage workers, who comprise one third of all workers in the U.S. and are essential to many industries, are more likely to be physically inactive and to have cardiometabolic conditions and depression, yet the participants are half as likely as higher wage workers to utilize preventive care. Targeted workplace initiatives have been successful in improving employee health, but low-wage workers are difficult to engage, in part due to a high burden of social disadvantage (e.g., food and housing insecurity, time and financial constraints). There are few, if any, workplace interventions for depression that specifically target low-wage workers and the participants unique social risk factors. This study was designed using a planned adaptation approach that involved low-wage workers in the design of the intervention to increase engagement and feasibility. The study will test an evidence-based 8-session telephone-delivered depression intervention for working adults, Be Well at Work, and critical adaptations for low-wage workers: assessment and referrals for social determinants of health (e.g., food and housing insecurity, financial stress), physical activity promotion, and personalized text message behavioral support. The adapted intervention, Be Well at Work-PLUS, will be evaluated through a pilot randomized controlled trial comparing Be Well at Work-PLUS to a waitlist condition. The primary objectives are to assess acceptability, feasibility, and preliminary clinical outcomes. The primary preliminary clinical outcome is depression symptom severity, and secondary outcomes are physical activity, sleep quality, blood pressure, and BMI).

ELIGIBILITY:
Inclusion Criteria:

* part-time or full-time employment (at least 20 hours per week);
* ≥18 years old;
* employed in low-wage-earning jobs in the Environmental Services or Food & Nutrition Services Departments;
* presence of depression symptoms as measured by the Patient Health Questionnaire-9 item version; individuals who score ≥5 (indicating mild depression symptoms or higher) will be eligible;
* presence of impairment in work functioning, as measured by the Work Limitations Questionnaire; individuals who score ≥5% (indicating mild work productivity loss) will be eligible;
* possession of a cell phone with ability to receive text-messages;
* Fluent in either English or Spanish.

Exclusion Criteria:

* plan to leave Scripps employment in <6 months;
* severe mental illness or substance use condition (e.g., bipolar disorder, schizophrenia, active alcohol use disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Intervention feasibility | From enrollment to end of treatment (approximately 4 months after enrollment).
  Feasibility will be assessed by the number of intervention sessions completed. The intervention will be considered feasible if the majority of participants complete 75% (6 of 8) or more phone sessions.
Depression symptoms | From baseline through end of treatment (approximately 4 months after enrollment).
  Depression symptoms will be measured with the Patient Health Questionnaire - 9 item version (range 0-27, higher = worse depression symptoms)

SECONDARY OUTCOMES:
Work limitations | From baseline to end of treatment (approximately 4 months after enrollment)
  Work limitations (range: 0-100%, higher = more limitation) will be measured by the Work Limitations Questionnaire.
Perceived stress | From baseline to end of treatment (approximately 4 months after enrollment)
  Perceived stress measured by the Perceived Stress Scale (range 0-40, higher = more perceived stress).
Sleep quality | Baseline, follow-up (4 months)
  Sleep quality and duration as measured by the Pittsburgh Sleep Quality Index (range: 0-21, higher scores indicate worse sleep quality).
Physical activity - step count | Baseline, follow-up (4 months)
  Weekly step count as measured by wrist-worn FitBit watch
Body Mass Index | Baseline, follow-up (4 months)
  A weight-to-height ratio, calculated by dividing participant's weight in kilograms by height in meters squared.
Blood pressure | Baseline, Follow-up (4 months)
  Resting systolic and diastolic blood pressures
Physical Activity (self-report) | Baseline, Follow-up (4 months)
  Self-reported physical activity using the Global Physical Activity Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L McCurley, PhD MPH, Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Currently we do not plan to share data as this is an open pilot study with a small number of participants (N=60), and thus it could be possible identify individuals.